CLINICAL TRIAL: NCT07139444
Title: Use of Physical Therapy Outcome Measures to Predict Discharge Destination in People With Stroke From Acute Care Hospital
Status: Not yet recruiting | Type: Observational
Sponsor: New York Presbyterian Brooklyn Methodist Hospital (Other)
Collaborators: Nova Southeastern University (Other)
Responsible Party: Principal Investigator, Aniketh Chavan, Physical Therapist, New York Presbyterian Brooklyn Methodist Hospital
Other Study IDs: 2143128-1
Record Dates: First submitted 2025-08-17; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Stroke, Acute; Cerebrovascular Accident; Stroke; Stroke Hemorrhagic
Keywords: stroke; PASS; AM-PAC "6-Clicks"; MSAS; acute care hospital; physical therapy outcome measures
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: One time Physical Therapy Evaluation — A physical therapist will perform an evaluation which will consist of history taking and assessing the following: strength, endurance, range of motion, sitting/standing balance, sensory testing, and skin integrity. Following these assessments, the physical therapist will assess participant's functional mobility which involves assessing how you get out of bed, standing up, and walking. The physical therapist will also assess the participant on three tests which help determine your balance and assistance required with functional mobility. The tests that will be performed in no particular order are PASS, MSAS, AM-PAC "6-Clicks", OPS, MRS, and FCI. Data for the AM-PAC daily activity and applied cognition domains will be obtained from the patient's chart from the Occupational Therapy evaluation. Discharge destination information will be obtained from the PT evaluation and the discharge destinations will be acute/inpatient rehab, SAR, SNF, Home with or without home PT, and outpatient PT.

SUMMARY:
Physical therapy assessments assist in discharge planning along with demographic and social factors for patients with stroke in acute care. Understanding where a patient can be discharged to, based on the patient's functional status post stroke is important to be able to use resources effectively, decrease length of stay, and facilitate early initiation of rehabilitation services if needed. Standardized outcome measures can help quantify functional deficits and the scores on the standardized outcome measures can in turn guide the discharge planning process. The Activity Measure for Post Acute Care "6-Clicks" (AM-PAC "6-Clicks") has been used in the acute care setting to guide discharge planning. Based on its cutoff scores, it also can assist in predicting discharge destination. The Mobility Scale for Acute Stroke (MSAS) has been used to determine discharge to home versus not home in patients with stroke. Understanding the validity of the MSAS in comparison with the Postural Assessment Scale for Stroke (PASS) and the AM-PAC "6-Clicks" can be beneficial as the MSAS is a stroke specific outcome measure which is mainly used in acute care and is easy to administer. It can be administered in a short duration and consists of mobility and balance assessments which can help determine functional deficits.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who have a confirmed diagnosis of a first acute, single or multiple infarct, ischemic or hemorrhagic in nature by imaging.
2. Individuals who are 18 years of age or older.
3. Individuals must be non-institutionalized prior to hospital admission.
4. Individuals whose primary spoken and written language is English.
5. Individuals who are referred for physical therapy in acute care.

Exclusion Criteria:

1. Individuals who are non-ambulatory prior to hospital admission.
2. Individuals having a diagnosis of secondary major trauma or subarachnoid hemorrhage.
3. Individuals with any comorbidity that prevents him/her from completing the tests such as a previous neurological injury or recent orthopedic diagnoses.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of interest is individuals with acute stroke admitted to the neurology unit of New York Presbyterian Brooklyn Methodist hospital in New York. 532 patients with stroke were admitted to the hospital in the year 2022. Participants will be recruited based on a sample of convenience. All people with a diagnosis of stroke admitted to the neurology unit of the acute care hospital will be screened for participation using the medical record. Patients with stroke who meet the inclusion criteria will be offered the opportunity to participate in the research study. Patients who agree to participate will be provided with an informed consent form which will be signed by the patient or health care proxy. If a patient chooses not to participate in the study, the patient will still receive physical therapy services similar to the study participant.
Sampling Method: Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2025-09 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Mobility Scale for Acute Stroke (MSAS) | Baseline
  The MSAS is a six-item scale which consists of components that are routinely assessed in patients by physical therapists. The components are bridging, sit from supine and then return to supine, sitting balance to be held for 3 minutes, sit to stand from a chair without using arms, standing balance for 1 minute, and gait testing for 10 m with or without an assistive device. The scores for each domain range from 6 to 36. The cut off score is 26 with scores above 26 indicating possible discharge to home and below 26 indicating need for institutionalization.
Postural Assessment Scale for Stroke (PASS) | Baseline
  The PASS consists of 12-items assessing balance ability to maintain postures or while changing postures. The score range for the PASS is 0 to 36 with lower scores indicating greater balance impairments. The 12 items consist of sitting without support, standing with support, standing without support, standing on nonparetic leg, standing on paretic leg, supine to paretic side lateral, supine to nonparetic side lateral, supine to sitting up on edge of the mat, sitting on the edge of the mat to supine, sitting to standing up, standing up to sitting down, and standing - picking up a pencil from the floor.
Activity Measure for Post-Acute Care "6-Clicks" (AM-PAC "6-Clicks") | Baseline
  The AM-PAC was developed to assess activity level post-acute care. It consists of three domains - basic mobility, daily activity, and applied cognition and each of the three domains consists of six items. The raw scores for each domain range from 6 to 24. A higher raw score indicates less functional limitations. The cutoff score for medically complex patients is 42.9 for the basic mobility domain and 39.4 for the daily activity domain.

SECONDARY OUTCOMES:
Orpington Prognostic Scale (OPS) | Baseline
  The OPS consists of four domains namely deficits in upper extremity strength, upper extremity proprioception, balance, and cognition. The total score consists of adding all four domains together along with 1.6. The total score can range from 1.6 to 6.8. The cutoff scores range from < 3.2 to > 5.2, where < 3.2 indicates a high likelihood of discharge home; a score between 3.2 and 5.2 respond better to inpatient rehabilitation; and a score of > 5.2 indicates increased risk of institutionalization as patients are typically dependent.
Modified Rankin Scale (MRS) | Baseline
  The MRS is a global outcomes rating scale which ranges from 0 (no impairment) to 5 (severe disability- patient is bedridden, incontinent, and requires constant nursing care and attention) and 6 (death). A higher score indicates greater impairment.
Functional Comorbidity Index (FCI) | Baseline
  The FCI was developed to assess comorbidity and used physical function as the outcome. It consists of an 18-item list of diagnoses. The scores range from 0 to 18 which is the cumulative sum of the comorbidities present.

CONTACTS AND LOCATIONS:
Overall Officials: Asad Siddiqi, DO, Principal Investigator — New York Presbyterian Brooklyn Methodist Hospital
Locations (1):
- New York Presbyterian Brooklyn Methodist Hospital, Brooklyn, New York, United States

IPD SHARING:
Plan to Share IPD: No
The data will be deidentified and will be saved on a password protected drive. In addition, only personnel who are associated with the study will have access to the study specific records in the database. For any adverse events that happen during the physical therapy assessment, they will be documented, and the medical team will be notified. A data transfer usage agreement will be established between Nova Southeastern University and New York Presbyterian Brooklyn Methodist Hospital.